CLINICAL TRIAL: NCT05825833
Title: Infliximab Efficacy in Relation to Therapeutic Drug Monitoring and Serum Tumor Necrosis Factor (TNF)α Levels in Pediatric Hematopoietic Stem Cell Transplant Recipients
Brief Title: Infliximab Efficacy in Relation to Therapeutic Drug Monitoring and Serum TNFα Levels in Pediatric HSCT
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 18/22
Record Dates: First submitted 2023-03-29; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Acute Graft-versus-host Disease
Keywords: Acute graft-versus-host disease; Infliximab; TNFα; Hematopoietic Stem Cell Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite significant progress in overall survival and event-free survival in Pediatric Hematopoietic Stem Cell Transplant (HSCT), therapeutic options for graft-versus-host disease control remain limited, particularly in steroid-refractory patients. Several strategies have been proposed in the last 20 years but so far, the results have been inconclusive, complicated by the small population afflicted, inconsistent treatment schedules, different disease classifications and diagnosis methods. The number of studies concerning pediatric patients are even smaller. First line therapy for acute graft-versus-host disease (aGVHD) is steroid treatment that achieve partial or complete remission of the disease in a variable percentage of cases (40-60%), depending mainly to severity of GVHD and number of organ involvement, with hepatic and gastrointestinal GVHD particularly refractory to steroid treatment. For second line therapy there is no a standardized strategy with a great variety of immunosuppressive treatment without a real superiority of a drug in comparison to another. Steroid refractory acute GVHD is therefore one of the most important challenges in HSCT field. One of the more promising routes, based on published data and clinical experience, is the off-label use of Infliximab, an anti-Tumor Necrosis Factor α drug (already approved for many rheumatologic and autoimmune diseases) administered as a second line treatment in patients with steroid-refractory aGVHD at the standardized dosage of 10 mg/kg, although limited evidence has been published to validate this subscription. Biological pattern that could explain susceptibly of GVHD to infliximab treatment could lie in physiopathology of acute gastrointestinal GVHD that may resemble ulcerative rectocolitis. In this case, relation to Therapeutic Drug Monitoring (TDM) and Tumor Necrosis Factor α (TNFα) levels could be critical in monitoring the efficacy of the drug and need of further doses. Limited published data and clinical experience show that Infliximab may be able to further control symptoms and inflammatory response in a promising percentage of treated patients, although some have no benefit from the treatment. The aim of this study is to analyze the role of TNFα concentration in aGVHD, its levels fluctuation and clinical response of GVHD to Infliximab treatment in steroid-refractory pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients between 0 and 18;
* Allogeneic HSCT recipient;
* Onset of clinical signs of acute skin, gastrointestinal or hepatic GVHD according to the Glucksberg classification;
* At least five days of steroid treatment (minimum 1 mg/kg of methylprednisone or equivalent) for systemic aGVHD without clinical or laboratory signs of response or no steroid treatment for onset of grade I-II hepatic/gastroesophageal/intestinal isolated aGVHD;
* Patients who consent for the off-label use of infliximab and data processing for research purposes;
* At least one dose of infliximab received during aGVHD management;
* Minimum follow-up after infliximab administration of 6 months

Exclusion Criteria:

* Active fungal or bacterial infection with life-threatening clinical condition (shock or respiratory distress needing mechanical ventilation)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with steroid-refractory aGVHD and treated with infliximab
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between TNFα plasmatic concentration and serum infliximab levels | At day 56 after starting infliximab treatment
  TNFα levels and infliximab concentration will be measured in peripheral blood sample (serum)

SECONDARY OUTCOMES:
Correlation between TNFα concentration and serum infliximab levels | At day 7 after starting infliximab treatment
  TNFα levels and infliximab concentration will be measured in peripheral blood sample (serum)
Association between Baseline TNFα concentration and aGVHD overall severity | Before starting infliximab treatment
  TNFα levels will be measured in peripheral blood sample (serum)
Number of patients who achieved a significant drop of TNFα concentration after infliximab treatment | At day 7 after starting infliximab treatment
  TNFα levels will be measured in peripheral blood sample (serum)
Number of patients who achieved a significant drop of TNFα concentration after infliximab treatment | At day 14 after starting infliximab treatment
  TNFα levels will be measured in peripheral blood sample (serum)
Number of patients who achieved a significant drop of TNFα concentration after infliximab treatment | At day 28 after starting infliximab treatment
  TNFα levels will be measured in peripheral blood sample (serum)
Number of patients who achieved a significant drop of TNFα concentration after infliximab treatment | At day 42 after starting infliximab treatment
  TNFα levels will be measured in peripheral blood sample (serum)
Number of patients who achieved a significant drop of TNFα concentration after infliximab treatment | At day 56 after starting infliximab treatment
  TNFα levels will be measured in peripheral blood sample (serum)
Response to infliximab treatment for aGVHD | At day 7 after starting infliximab treatment
  Number of patients who had Complete Response (CR), Partial Response (PR) or Non-Response (NR). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Response to infliximab treatment for aGVHD | At day 14 after starting infliximab treatment
  Number of patients who had Complete Response (CR), Partial Response (PR) or Non-Response (NR). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Response to infliximab treatment for aGVHD | At day 28 after starting infliximab treatment
  Number of patients who had Complete Response (CR), Partial Response (PR) or Non-Response (NR). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Response to infliximab treatment for aGVHD | At day 42 after starting infliximab treatment
  Number of patients who had Complete Response (CR), Partial Response (PR) or Non-Response (NR). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Response to infliximab treatment for aGVHD | At day 56 after starting infliximab treatment
  Number of patients who had Complete Response (CR), Partial Response (PR) or Non-Response (NR). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Infliximab serum concentration in patients with clinical CR, PR, NR. | At day 7 after starting infliximab treatment
  Infliximab concentration will be measured in peripheral blood sample (serum). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Infliximab serum concentration in patients with clinical CR, PR, NR. | At day 14 after starting infliximab treatment
  Infliximab concentration will be measured in peripheral blood sample (serum). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Infliximab serum concentration in patients with clinical CR, PR, NR. | At day 28 after starting infliximab treatment
  Infliximab concentration will be measured in peripheral blood sample (serum). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Infliximab serum concentration in patients with clinical CR, PR, NR. | At day 42 after starting infliximab treatment
  Infliximab concentration will be measured in peripheral blood sample (serum). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Infliximab serum concentration in patients with clinical CR, PR, NR. | At day 56 after starting infliximab treatment
  Infliximab concentration will be measured in peripheral blood sample (serum). Response is defined as complete resolution of GVHD symptoms and normalization of the biochemical parameters of inflammation.
Percentage of infection during follow-up | At 6 months after starting infliximab treatment
  Viral reactivation (Cytomegalovirus and Epstein-Barr virus), bacterial and fungal infection will be evaluated by medical records
Percentage of infection during follow-up | At 12 months after starting infliximab treatment
  Viral reactivation (Cytomegalovirus and Epstein-Barr virus), bacterial and fungal infection will be evaluated by medical records
Percentage of chronic GVHD | At 6 months after starting infliximab treatment
  Evaluated by medical records
Percentage of chronic GVHD | At 12 months after starting infliximab treatment
  Evaluated by medical records
Percentage of relapse | At 6 months after starting infliximab treatment
  Evaluated by medical records
Percentage of relapse | At 12 months after starting infliximab treatment
  Evaluated by medical records
Transplant-related mortality | At 6 months after starting infliximab treatment
  Evaluated by medical records
Overall survival | At 6 months after starting infliximab treatment
  Evaluated by medical records
Transplant-related mortality | At 12 months after starting infliximab treatment
  Evaluated by medical records
Overall survival | At 12 months after starting infliximab treatment
  Evaluated by medical records

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Maestro, PharmD, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy